CLINICAL TRIAL: NCT03493191
Title: A Phase I, Randomized, Double-blind, Placebo-Controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous SHR0410 in Healthy Male Participants
Brief Title: A Single Dose Study of SHR0410 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Collaborators: Linear Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR0410-101-AU
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0.5 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 0.5μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 0.5μg/kg SHR0410
- 1 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 1μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 1μg/kg SHR0410
- 2 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 2μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 2μg/kg SHR0410
- 5 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 5μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 5μg/kg SHR0410
- 10 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 10μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 10μg/kg SHR0410
- 20 μg/kg SHR0410 (Experimental): 8 subjects will be randomized in a 3:1 ratio to receive a single dose of either 10μg/kg SHR0410 (n=6) or placebo (n=2)
  Interventions: Drug: 20μg/kg SHR0410

INTERVENTIONS:
Drug: 0.5μg/kg SHR0410 — a single dose of 0.5μg/kg SHR0410
  Arms: 0.5 μg/kg SHR0410
Drug: 1μg/kg SHR0410 — a single dose of 2μg/kg SHR0410
  Arms: 1 μg/kg SHR0410
Drug: 2μg/kg SHR0410 — a single dose of 2μg/kg SHR0410
  Arms: 2 μg/kg SHR0410
Drug: 5μg/kg SHR0410 — a single dose of 5μg/kg SHR0410
  Arms: 5 μg/kg SHR0410
Drug: 10μg/kg SHR0410 — a single dose of 10μg/kg SHR0410
  Arms: 10 μg/kg SHR0410
Drug: 20μg/kg SHR0410 — a single dose of 20μg/kg SHR0410
  Arms: 20 μg/kg SHR0410

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending-dose study to investigate the effect of a single intravenous (IV) dose of SHR0410 at 6 dose levels (0.5 μg/kg, 1 μg/kg, 2 μg/kg, 5 μg/kg, 10 μg/kg and 20 μg/kg) in healthy participants.

DETAILED DESCRIPTION:
Forty eight eligible participants will be enrolled into the 6 dose cohorts. For each cohort, a sentinel group of 2 subjects (1 receiving SHR0410 and 1 receiving placebo) will be dosed first (1:1 ratio). If no drug related adverse events occur in the sentinel participants, the remaining 6 subjects in a cohort will be dosed on the next day or later in a 5:1 ratio (5 subjects receiving SHR0410 and 1 subject receiving placebo). SHR0410 will be diluted in saline and administered as a 15 min constant dose IV infusion at a rate of 20 ml/hr on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Male between the ages of 18 and 45 years, inclusive.
2. Body mass index (BMI) of 18.0 to 30.0 kg/m2 and a total body weight of 50 kg to 125kg, inclusive.
3. Considered generally healthy upon completion of medical history, physical examination, vital signs, SpO2, laboratory parameters, and ECG, as judged by the Investigator.

Exclusion Criteria:

1. Known sensitivity to any of the components of the investigational product formulation, or any other opioids.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
3. Any other medical or psychological condition, which in the opinion of the Investigator, might create undue risk to the participant or interfere with the participant's ability to comply with the protocol requirements, or to complete the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events in terms of changes in Hematology | Up to Day 8
  Hemoglobin Hematocrit Erythrocytes count Mean cell volume, Mean cell hemoglobin concentration, Leukocytes count, Neutrophils count, Lymphocytes count, Monocytes count, Eosinophils count, Basophils count, Platelets count
Incidence of Adverse events in terms of changes in Urinalysis | Up to Day 8
  Urobilinogen Dipstick urinalysis, including: pH, Specific gravity, Protein, Blood, Leukocytes, Glucose, Ketones, Bilirubin, Nitrites
Incidence of Adverse events in terms of changes in Biochemistry (fasting) | Up to Day 8
  Including Serum creatinine, Urea, Alanine aminotransferase, Aspartate aminotransferase, Gamma glutamyl transferase, Total bilirubin, Total protein, Albumin, Alkaline phosphatase, Serum uric acid, Glucose, Triglycerides, Total cholesterol, High-density lipoprotein cholesterol, Low-density lipoprotein cholesterol
Incidence of Adverse events in terms of changes in Physical examinations | Up to Day 8
  Review of body weight and height; general appearance; head; eyes; ears/nose/throat; neck; lymph nodes; neurological and musculoskeletal systems; heart; lungs; abdomen; skin; and extremities
Incidence of Adverse events in terms of changes in Vital signs | Up to Day 8
  Oral temperature, respiratory rate, blood pressure, and pulse rate
Incidence of Adverse events in terms of changes in 12-lead ECGs | Up to Day 8
  The 12-lead ECGs must be recorded after the subjects have rested in the supine position for 5 minutes to ensure a stable baseline.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 24 hours post dose
  Plasma SHR0410 Area Under the Concentration-time Curve (AUC)
Time to the peak plasma concentration (Tmax) | Up to 24 hours post dose
  Time to Maximum Plasma SHR0410 Concentration
Peak Plasma Concentration (Cmax) | Up to 24 hours post dose
  Peak Plasma SHR0410 Concentration
Half-time (T1/2) | Up to 24 hours post dose
  Half-time of SHR0410
Urine output rate | Up to 48 hours post dose
  Changes in urine output rate from baseline
Serum prolactin release rate | Up to 48 hours post dose
  Changes in serum prolactin release rate from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Limited, Nedlands, Australia